CLINICAL TRIAL: NCT04607434
Title: Mechanism of Delayed Neutrophil Apoptosis in Acute Lung Injury: Effects of Ginsenoside Derivatives on the Improvement of Delayed Neutrophil Apoptosis
Brief Title: Mechanism of Delayed Neutrophil Apoptosis in Acute Lung Injury
Status: Completed | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Zhongmin Liu, Director of critical care medicine center, The First Hospital of Jilin University
Other Study IDs: jdyyicu3
Record Dates: First submitted 2020-10-26; First posted 2020-10-29 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Acute Lung Injury/Acute Respiratory Distress Syndrome (ARDS); Neutrophils; Apoptosis; Immunosuppression; Pathogenesis
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The peripheral blood of the patient was centrifuged and the supernatant was reserved for cryopreservation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ocotillol Type Ginsenoside Derivatives — Peripheral blood PMN of patients with ARDS were taken. The neutrophils isolated from peripheral blood of ARDS patients were incubated with different doses of OCT glycine derivatives (20,50,100 UM) for 20 h

SUMMARY:
Literature basis Acute respiratory distress syndrome (ARDS) is a clinical syndrome characterized by respiratory distress and progressive hypoxemia, which is caused by diffuse alveolar and pulmonary interstitial edema caused by various pulmonary and extrapulmonary factors other than cardiogenic factors. ARDS incidence rate is as high as 75 /10 000 per year, and sepsis and pulmonary infection are the most common causes. In the past, it was generally believed that excessive immune activation is the core of the pathophysiology of ARDS, and neutrophils are recognized as the core driver of inflammatory hyperactivity and lung injury in ARDS. Although some progress has been made in the epidemiology, pathogenesis and pathophysiology of ARDS in the past 50 years, and the clinical outcomes of some patients with ARDS have been improved by optimizing the mode of mechanical ventilation and fluid treatment, as well as prone ventilation and the use of muscle relaxants, ARDS is still one of the most common causes of death and disability in intensive care units, The mortality rate of the disease is currently as high as 30-40%. There is still a lack of effective drugs for the treatment of ARDS in clinic, and even glucocorticoids applied for immune overactivation have not achieved good results. This is related to the unclear pathogenesis of ARDS. Therefore, it is still a hot and difficult point to further explore the pathogenesis and progression of ARDS and find new therapeutic targets.

In the past, mature PMN in peripheral blood was generally considered as a functional cell in the end stage, but it is widely involved in different innate immune responses (including inflammation, infection, tumor, autoimmunity, etc.) and can adopt very different effector mechanisms. Therefore, with the deepening of research, neutrophil subtypes with different functions (such as immune regulation and repair) have been identified in recent years: cd16dimcd62lbrightpmn and cd16brightcd62ldimmpmn. In the steady state of healthy people, the classic mature neutrophils (cd16brightcd62lbright) in peripheral blood account for more than 98% of the total PMN, and the proportion of the two neutrophil subtypes is relatively low. In the inflammatory state, the proportion of cd16dimcd62lbright and cd16brightcd62ldim neutrophils increased significantly. Proteomic analysis showed that there were significant differences between the two subtypes of neutrophils. The nucleus of cd16dimcd62lbright neutrophil subgroup is banded, which is released from bone marrow after being stimulated by lipopolysaccharide (LPS). It accounts for 20% - 25% of PMN in whole blood in LPS infection model. The apoptosis rate is significantly reduced, and the bacteriostatic effects such as oxidative burst and phagocytosis are significantly enhanced; On the contrary, cd16brightcd62ldim neutrophil subgroup has reduced antibacterial ability and shows immunosuppressive phenotype. It is a newly discovered neutrophil subtype with immunosuppressive function in recent years, which can inhibit T cell proliferation, which is related to immunosuppression in the experimental human endotoxemia model.

In our previous studies, we have successfully obtained a new amino acid derivative of ocotillol ginsenoside, which may have the pharmacological activities of ocotillol ginsenoside and glycine, and has a potential role in improving the delay of apoptosis and immunosuppression of ARDS neutrophil subtypes, and has the potential of new drug development for the treatment of ARDS.

The experimental steps are as follows:

Firstly, the peripheral blood of ARDS patients in ICU was collected, and neutrophils were isolated from the peripheral blood. The proportion of neutrophil subtypes and the degree of apoptosis were detected by flow cytometry. Co culture with human T lymphocytes in vitro to observe its ability to inhibit T cell proliferation. Then, the neutrophils of ARDS patients were cultured with different doses of ginsenoside glycine derivatives, and the detection of the above indexes was repeated again. Finally, the mechanism of neutrophils in the pathogenesis and progression of ARDS was discussed.

DETAILED DESCRIPTION:
1. Literature basis cute respiratory distress syndrome (ARDS) is a clinical syndrome characterized by respiratory distress and progressive hypoxemia, which is caused by diffuse alveolar and pulmonary interstitial edema caused by various pulmonary and extrapulmonary factors other than cardiogenic factors. ARDS incidence rate is as high as 75 /10 000 per year, and sepsis and pulmonary infection are the most common causes. In the past, it was generally believed that excessive immune activation is the core of the pathophysiology of ARDS, and neutrophils are recognized as the core driver of inflammatory hyperactivity and lung injury in ARDS. Although some progress has been made in the epidemiology, pathogenesis and pathophysiology of ARDS in the past 50 years, and the clinical outcomes of some patients with ARDS have been improved by optimizing the mode of mechanical ventilation and fluid treatment, as well as prone ventilation and the use of muscle relaxants, ARDS is still one of the most common causes of death and disability in intensive care units, The mortality rate of the disease is currently as high as 30-40%. There is still a lack of effective drugs for the treatment of ARDS in clinic, and even glucocorticoids applied for immune overactivation have not achieved good results. This is related to the unclear pathogenesis of ARDS. Therefore, it is still a hot and difficult point to further explore the pathogenesis and progression of ARDS and find new therapeutic targets.

In the past, mature PMN in peripheral blood was generally considered as a functional cell in the end stage, but it is widely involved in different innate immune responses (including inflammation, infection, tumor, autoimmunity, etc.) and can adopt very different effector mechanisms. Therefore, with the deepening of research, neutrophil subtypes with different functions (such as immune regulation and repair) have been identified in recent years: cd16dimcd62lbrightpmn and cd16brightcd62ldimmpmn. In the steady state of healthy people, the classic mature neutrophils (cd16brightcd62lbright) in peripheral blood account for more than 98% of the total PMN, and the proportion of the two neutrophil subtypes is relatively low. In the inflammatory state, the proportion of cd16dimcd62lbright and cd16brightcd62ldim neutrophils increased significantly. Proteomic analysis showed that there were significant differences between the two subtypes of neutrophils. The nucleus of cd16dimcd62lbright neutrophil subgroup is banded, which is released from bone marrow after being stimulated by lipopolysaccharide (LPS). It accounts for 20% - 25% of PMN in whole blood in LPS infection model. The apoptosis rate is significantly reduced, and the bacteriostatic effects such as oxidative burst and phagocytosis are significantly enhanced; On the contrary, cd16brightcd62ldim neutrophil subgroup has reduced antibacterial ability and shows immunosuppressive phenotype. It is a newly discovered neutrophil subtype with immunosuppressive function in recent years, which can inhibit T cell proliferation, which is related to immunosuppression in the experimental human endotoxemia model.

In our previous studies, we have successfully obtained a new amino acid derivative of ocotillol ginsenoside, which may have the pharmacological activities of ocotillol ginsenoside and glycine, and has a potential role in improving the delay of apoptosis and immunosuppression of ARDS neutrophil subtypes, and has the potential of new drug development for the treatment of ARDS.

2. The experimental steps are as follows:

1. Peripheral blood samples from patients with ARDS were collected to detect inflammatory markers;
2. Neutrophils were isolated from peripheral blood of patients with ARDS;
3. The proportion of neutrophil subtypes was detected by flow cytometry, and the neutrophil subtypes were isolated;
4. Neutrophil subtypes were co cultured with peripheral blood T lymphocytes to detect their ability to inhibit T cell proliferation and the apoptosis of neutrophil subtypes;
5. Peripheral blood neutrophils and different doses of ginsenoside glycine derivatives in patients with ARDS (2050100 μ m) After incubation for 20h, the apoptosis rate was 28h.
6. Bax, Mcl-1 and cleaved caspase-3 were detected by Western blot.
7. High throughput PCR and mapp-4 were used to detect the expression of apoptosis related genes in akg38k pathway.
8. Metabolomic analysis: collect the peripheral blood of ARDS patients for metabolomic analysis.

3. Research methods

1. Diagnostic criteria: refer to the 2012 Berlin standard for the diagnostic criteria of ARDS.
2. Inclusion criteria: (1) age ≥ 18 years old; (2) Diagnosis of acute lung injury within 24 hours (Berlin diagnostic criteria for acute lung injury)
3. Exclusion criteria: (1) age < 18 years; (2) Discharge or death within 48 hours after admission; (3) Pregnancy or puerperium; (4) Patients with immunosuppression.

4. Test procedure

1. Methods: ICU patients who met the inclusion criteria were selected
2. Informed consent process: sign the informed consent form after communicating with the patient or legal representative

5. Start and end of the experiment Informed consent was signed in January 2020

6. Data security and monitoring plan The patient's medical records (study medical records / CRF, test forms, etc.) will be kept completely in the hospital. The doctor will record the results of laboratory tests and other examinations in his medical record. The researchers, the ethics committee and the drug administration will be allowed access to his medical records. No public report on the results of the study will reveal the individual identity of the patient. We will make every effort to protect patient information to the extent permitted by law. According to medical research ethics, except for personal privacy information, experimental data will be available for public inquiry and sharing, and the query and sharing will be limited to the electronic database based on the network to ensure that no personal privacy information will be disclosed.

7. Abide by ethical principles and relevant laws and regulations Whether or not to participate in the study depends entirely on the wishes of patients and their legal representatives. Patients and their families may refuse to participate in the study or withdraw from the study at any time during the course of the study. This will not affect the relationship between the patient and his doctor, nor will it affect the loss of medical or other benefits for the patient.

8. Statistical analysis plan SPSS15.0 software was used for statistical analysis. The measurement data were expressed as mean ± standard deviation, t test or nonparametric test was used for comparison between groups, chi square test was used for counting data, and linear correlation analysis was used for the relationship between variables, P < 0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion criteria:

* 90≥age ≥ 18 years old
* patients in ICU; within 24 hours of diagnosis of acute lung injury (Berlin criteria for acute lung injury)

Exclusion criteria:

* death within 48 hours of admission
* Pregnancy or puerperium
* Patients with immunosuppression

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients admitted to the first hospital of Jilin University in Changchun City, Jilin Province, China
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Inpatient mortality rate | Within 28 days
  Inpatient mortality during ICU stay in the enrolled patients

SECONDARY OUTCOMES:
New infection rate | 5 days after check-in at ICU
  Incidence of new infections in ARDS patients after admission to ICU5 days
the apoptosis rate | 20 hours
  Peripheral blood neutrophils from patients with ARDS and healthy controls were incubated with different doses of OCT glycine derivatives (20, 50, 100 UM) for 20 h, and the apoptosis rate was measured

CONTACTS AND LOCATIONS:
Overall Officials: jing zhang, doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- first hospital of Jilin University, Changchun, China